CLINICAL TRIAL: NCT04099810
Title: Assessment of Right Ventricular Volume in Pediatric Patients - Is Apical or Subcostal Window More Accurate?
Brief Title: Assessment of Right Ventricular Volume in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David Harrild, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00033035
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Function
Keywords: three-dimensional echocardiography; right ventricular volumes; cardiac magnetic resonance
MeSH Terms: interventions — Echocardiography, Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients undergoing Cardiac MRI (Other): Patients scheduled to undergo cardiac magnetic resonance for clinical reason will be asked if they are willing to undergo additional non invasive testing (three-dimensional echocardiography) which will take about 15-20 minutes
  Interventions: Diagnostic Test: three-dimensional echocardiography

INTERVENTIONS:
Diagnostic Test: three-dimensional echocardiography — A focused echocardiographic exam will be performed. In details will be acquired:
  * high frame rate imaging clips acquired in a static position with attention to endocardial border optimization, minimum of 3 beats recorded with 'Acquire 2', of: a. Left ventricle 2c/3c/4c; b. left ventricle SAB, SAX-M, SAX-A; c. right ventricular focused apical view.
  * Full volumes: a. 3d left ventricular apical acquisition; b. right ventricular apical acquisition; c. subcostal right ventricular acquisition.

SUMMARY:
Most publication are basing RV volumes on images acquired from the apical window. However, some data have called the practice of basing these images on apical window into question. Moreover, despite our best efforts, we have been unable, in our laboratory to reliably visualize RV outflow from the apical view. Therefore, with an identified group of trained sonographers, we plan to conduct a head-to-head comparison of RV volumes acquired from these two windows (apical and subcostal), with comparison to gold-standard CMR.

DETAILED DESCRIPTION:
The knowledge of right ventricular (RV) volumes is important from a clinical prospective. Traditionally, these volumes have been measured by cardiac magnetic resonance (CMR) because of its accuracy, reproducibility, and freedom from geometric assumptions. More and more, however, 3D echo has been used for assessment of ventricular volumes, first for left ventricle, now increasingly for RV. Most publication are basing RV volumes on images acquired from the apical window. However, some data have called the practice of basing these images on apical window into question. Moreover, despite our best efforts, we have been unable, in our laboratory to reliably visualize RV outflow from the apical view. An alternative view that can be used for RV 3D volume acquisition (first pioneered at BCH) is the subcostal view. Therefore, we plan to conduct a head-to-head comparison of RV volumes acquired from these two windows (apical and subcostal), with comparison to gold-standard CMR.

Hypothesis: RVEDV measured by the subcostal window is more accurate than RV volume measured in the apical window in a cohort of pediatric patients.

Analytic plan: Echocardiograms will be performed on the same day as the CMR, and will be performed by a group of sonographers trained in 3D volume acquisition. Descriptive statistics will include mean and median absolute % error and coefficients of variation. A paired t-test will be used to compare raw differences in %error for apical vs. subcostal window measurements. If the %error is highly skewed, a Wilcoxon signed-rank test will be used or the %error values will be log-transformed before application of the paired t-test (if no zero %error values exist). Linear regression will be used to estimate the window-differences in %error or log(%error) controlling for age and/or sedation status. Assessments of feasibility for both windows will be performed as described by Renella et al; and reproducibility of measurements made with echo vs. CMR will be also be graphically assessed using Bland-Altman plots of the raw measurements for data derived from each window. As a secondary (stratified) analysis, we anticipate dividing the cohort into 2 groups of 25 patients each (25 < 10y; 25 > 10y). Patients under 10y will typically be under anesthesia. Exploratory analyses will investigate subgroup differences defined by demographic/ surgical variables with respect to the magnitude of the difference between the 2 techniques. Of note the analyses performed above will also be performed for LV (in addition to RV) as a secondary analysis (with comparison of LV-specific vs. non-LV specific software, as appropriate).

Sample size/Power: funding is provided for 50 patients and this will be our target sample size. The analysis will be paired, to compare the %error (echo relative to MRI) measurements from apical vs. subcostal windows). To detect a 0.5 SD difference in apical vs. subcostal windows %error with 85% power, 38 subjects with echo & MRI are required. If the comparisons are performed stratified by age (25 subjects per age group), there is 80% power to detect a 0.58 SD difference in apical vs. subcostal windows %error.

Limitations: CMR, while considered a gold-standard, has a certain amount of intrinsic variability in volume measurement. Moreover, a statistically significant difference may not necessary be a clinically important difference. Patients will not have echo and CMR performed at the exact same time.

ELIGIBILITY:
Inclusion Criteria:

* Patients<18y scheduled to undergo CMR for clinical reasons.

Exclusion Criteria:

* Patients >18y

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mean absolute %error in end diastolic volume measurements | 0 days
  Mean absolute %error in end diastolic volume measurements (apical and subcostal windows) (echocardiographic vs. gold-standard CMR); echocardiographic right ventricular (RV) volumes measured using RV-specific software

SECONDARY OUTCOMES:
Mean absolute %error in right ventricular end systolic volume (RVESV) / right ventricular ejection fraction (RVEF) | 0 days
  Mean absolute %error in right ventricular end systolic volume (RVESV) / right ventricular ejection fraction (RVEF) (apical and subcostal windows) (echocardiographic vs. gold-standard cardiac MRI) for RV volumes measured using RV-specific software
Mean absolute %error in RVEDV/RVESV/RVEF (subcostal window) | 0 days
  Mean absolute %error in RVEDV/RVESV/RVEF (subcostal window) for RV volumes measured with RV nonspecific software vs. RV specific software

CONTACTS AND LOCATIONS:
Overall Officials: David M Harrild, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data has been considered until now.

REFERENCES:
- [Background] Kutty S, Zhou J, Gauvreau K, Trincado C, Powell AJ, Geva T. Regional dysfunction of the right ventricular outflow tract reduces the accuracy of Doppler tissue imaging assessment of global right ventricular systolic function in patients with repaired tetralogy of Fallot. J Am Soc Echocardiogr. 2011 Jun;24(6):637-43. doi: 10.1016/j.echo.2011.01.020. Epub 2011 Mar 9. PMID 21392939
- [Background] Geva T. Repaired tetralogy of Fallot: the roles of cardiovascular magnetic resonance in evaluating pathophysiology and for pulmonary valve replacement decision support. J Cardiovasc Magn Reson. 2011 Jan 20;13(1):9. doi: 10.1186/1532-429X-13-9. PMID 21251297
- [Background] Williams RG, Pearson GD, Barst RJ, Child JS, del Nido P, Gersony WM, Kuehl KS, Landzberg MJ, Myerson M, Neish SR, Sahn DJ, Verstappen A, Warnes CA, Webb CL; National Heart, Lung, and Blood Institute Working Group on research in adult congenital heart disease. Report of the National Heart, Lung, and Blood Institute Working Group on research in adult congenital heart disease. J Am Coll Cardiol. 2006 Feb 21;47(4):701-7. doi: 10.1016/j.jacc.2005.08.074. Epub 2006 Jan 26. PMID 16487831
- [Background] Oosterhof T, van Straten A, Vliegen HW, Meijboom FJ, van Dijk AP, Spijkerboer AM, Bouma BJ, Zwinderman AH, Hazekamp MG, de Roos A, Mulder BJ. Preoperative thresholds for pulmonary valve replacement in patients with corrected tetralogy of Fallot using cardiovascular magnetic resonance. Circulation. 2007 Jul 31;116(5):545-51. doi: 10.1161/CIRCULATIONAHA.106.659664. Epub 2007 Jul 9. PMID 17620511
- [Background] Knauth AL, Gauvreau K, Powell AJ, Landzberg MJ, Walsh EP, Lock JE, del Nido PJ, Geva T. Ventricular size and function assessed by cardiac MRI predict major adverse clinical outcomes late after tetralogy of Fallot repair. Heart. 2008 Feb;94(2):211-6. doi: 10.1136/hrt.2006.104745. Epub 2006 Nov 29. PMID 17135219
- [Background] Pennell DJ, Sechtem UP, Higgins CB, Manning WJ, Pohost GM, Rademakers FE, van Rossum AC, Shaw LJ, Yucel EK; Society for Cardiovascular Magnetic Resonance; Working Group on Cardiovascular Magnetic Resonance of the European Society of Cardiology. Clinical indications for cardiovascular magnetic resonance (CMR): Consensus Panel report. Eur Heart J. 2004 Nov;25(21):1940-65. doi: 10.1016/j.ehj.2004.06.040. No abstract available. PMID 15522474
- [Background] Kochav J, Simprini L, Weinsaft JW. Imaging of the right heart--CT and CMR. Echocardiography. 2015 Jan;32 Suppl 1:S53-68. doi: 10.1111/echo.12212. Epub 2014 Sep 19. PMID 25244072
- [Background] Monaghan MJ. Role of real time 3D echocardiography in evaluating the left ventricle. Heart. 2006 Jan;92(1):131-6. doi: 10.1136/hrt.2004.058388. No abstract available. PMID 16365369
- [Background] Aune E, Baekkevar M, Rodevand O, Otterstad JE. Reference values for left ventricular volumes with real-time 3-dimensional echocardiography. Scand Cardiovasc J. 2010 Feb;44(1):24-30. doi: 10.3109/14017430903114446. PMID 19626561
- [Background] Chahal NS, Lim TK, Jain P, Chambers JC, Kooner JS, Senior R. Population-based reference values for 3D echocardiographic LV volumes and ejection fraction. JACC Cardiovasc Imaging. 2012 Dec;5(12):1191-7. doi: 10.1016/j.jcmg.2012.07.014. PMID 23236967
- [Background] Muraru D, Badano LP, Peluso D, Dal Bianco L, Casablanca S, Kocabay G, Zoppellaro G, Iliceto S. Comprehensive analysis of left ventricular geometry and function by three-dimensional echocardiography in healthy adults. J Am Soc Echocardiogr. 2013 Jun;26(6):618-28. doi: 10.1016/j.echo.2013.03.014. Epub 2013 Apr 20. PMID 23611056
- [Background] Medvedofsky D, Addetia K, Patel AR, Sedlmeier A, Baumann R, Mor-Avi V, Lang RM. Novel Approach to Three-Dimensional Echocardiographic Quantification of Right Ventricular Volumes and Function from Focused Views. J Am Soc Echocardiogr. 2015 Oct;28(10):1222-31. doi: 10.1016/j.echo.2015.06.013. Epub 2015 Aug 1. PMID 26237996
- [Background] Ostenfeld E, Flachskampf FA. Assessment of right ventricular volumes and ejection fraction by echocardiography: from geometric approximations to realistic shapes. Echo Res Pract. 2015 Mar 1;2(1):R1-R11. doi: 10.1530/ERP-14-0077. Epub 2015 Jan 7. PMID 26693327
- [Background] Laser KT, Karabiyik A, Korperich H, Horst JP, Barth P, Kececioglu D, Burchert W, DallaPozza R, Herberg U. Validation and Reference Values for Three-Dimensional Echocardiographic Right Ventricular Volumetry in Children: A Multicenter Study. J Am Soc Echocardiogr. 2018 Sep;31(9):1050-1063. doi: 10.1016/j.echo.2018.03.010. Epub 2018 Jun 19. PMID 29908725
- [Background] Renella P, Marx GR, Zhou J, Gauvreau K, Geva T. Feasibility and reproducibility of three-dimensional echocardiographic assessment of right ventricular size and function in pediatric patients. J Am Soc Echocardiogr. 2014 Aug;27(8):903-10. doi: 10.1016/j.echo.2014.04.008. Epub 2014 May 14. PMID 24836600